CLINICAL TRIAL: NCT04979195
Title: Acute Kidney Injury Among COVID-19 Positive Patients is Associated With Higher Mortality: a Single-center Experience
Brief Title: Acute Kidney Injury Among COVID-19 Positive Patients
Acronym: AKI-COVID-19
Status: Completed | Type: Observational
Sponsor: Hamid Al-Essa Organ Transplant Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/1467
Record Dates: First submitted 2021-07-22; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-03

CONDITIONS: COVID-19 Positive Patients With Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients with stable renal function.
  Interventions: Other: Patients with stable normal kidney function; Other: Patients with unstable kidney function
- Group 2: Patients who developed AKI.
  Interventions: Other: Patients with stable normal kidney function; Other: Patients with unstable kidney function

INTERVENTIONS:
Other: Patients with stable normal kidney function — Covid-19 patients with stable kidney function will represent group 1.
  Other Names: Covid-19 patients with stable kidney fucntion.
Other: Patients with unstable kidney function — Covid-19 patients with unstable kidney function will represent group 2.
  Other Names: Covid-19 patients with unstable kidney fucntion.

SUMMARY:
In Kuwait, the total number of COVID-19 confirmed cases exceeds 5000 patients. Risk factors of possible risk factors of confirmed COVID-19 infection that developed major organ dysfunction are not yet identified among patients in Kuwait.

we aimed to describe the clinical characteristics of hospitalized symptomatic COVID-19 positive patients, assess possible risk factors of confirmed COVID-19 infection who developed major organ dysfunction, determine risk factors for renal dysfunction and their outcome and assess the response of critically ill patients to different therapeutic modalities.

DETAILED DESCRIPTION:
In this observational study, we will revise all medical records of hospitalized patients with laboratory-confirmed Covid-19, during the period between Feb till July 2020. A confirmed case of Covid-19 is defined as a positive result on high throughput sequencing or real-time reverse-transcriptase-polymerase-chain-reaction (RT-PCR) assay of nasal and pharyngeal swab specimens.12 We will include only laboratory-confirmed cases in the analysis.

We will extract patients' data with special stress on socio-demographic data, associated medical co-morbidities as diabetes, hypertension, ischemic heart disease, chronic lung disease, recent exposure history, clinical symptoms or signs of the upper and lower respiratory system, and laboratory findings on admission. Radiologic assessments will be included like chest radiography or computed tomography (CT), and all laboratory testing will be performed according to the clinical care needs of the patient.

We will determine the presence of a radiologic abnormality on the basis of the documentation or description in medical charts of infected patients; if imaging scans were available, they were reviewed by attending physicians in respiratory medicine who will extract the data. If a major disagreement between two reviewers happens it will be resolved by consultation with a third reviewer. Laboratory assessments will include a complete blood count, blood chemical analysis, coagulation testing, assessment of liver and renal function, and measures of electrolytes, C-reactive protein, procalcitonin, lactate dehydrogenase, creatine kinase, ferritin, D dimer, and troponin. The degree of severity of Covid-19 (severe vs. non-severe) at the time of admission will be defined using the American Thoracic Society guidelines for community-acquired pneumonia.

Data will be entered into a computerized database SPSS program file and cross-checked. If the core data are missing, requests for clarification will be sent to the coordinators, who subsequently will contact the attending clinicians.

Treatment and Complications:

We will report patients who are receiving antibiotics, antiviral (different regimens), those who required oxygen therapy (invasive, non-invasive ventilation or extracorporeal membrane oxygenation, (ECMO)), and those patients who received systemic steroid therapy. Moreover, the duration of hospitalization will be reported. Also, patients who developed acute kidney injury will be recorded and if they were dialyzed, all dialysis parameters will be recorded including any associated complications. All mortality patients will be reported with special stress on the cause of death.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients were included.
* Hospitalized with PCR confirmed COVID-19 infection.
* period between March to August 2020.

Exclusion Criteria:

* Pediatric patients Home isolated patients

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 649 COVID-19 positive patients were identified. Sixty-three were isolated at home and 586 cases needed hospital admission during the period between the 1st week of March till the end of August 2020. Among the hospitalized cases, 258 needed ICU care while 328 were managed in the COVID general wards. We compared patients with stable renal function (group 1, n=319) vs. those who developed AKI (group 2, n=267).
  We collected the data from COVID-19 positive patients that were diagnosed in all government hospitals in Kuwait. Clinical features, details of management, and both patient and renal outcomes were recorded. We compiled patients' data from the electronic database of the isolation hospitals where COVID -19 cases were managed. Approval for the study was obtained from the ethical committee of the Kuwait Ministry of Health.
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
patient survival | 30 days
  Patients who survived after 30 days.
Kidney survival | 30 days
  Patients who have stable basal kidney function.

CONTACTS AND LOCATIONS:
Locations (2):
- Kuwait (2):
  - Osama Gheith, Kuwait City, AZ
  - Osama Gheith, Kuwait City, Rf

IPD SHARING:
Plan to Share IPD: Undecided